CLINICAL TRIAL: NCT03274934
Title: The Effectiveness of the Novel Web- and Mobile-based Acceptance- and Commitment Therapy Program Youth COMPASS to Promote Adolescent Well-being and Life-control
Brief Title: The Effectiveness of the Mobile-based Youth COMPASS Program to Promote Adolescent Well-being and Life-control
Acronym: YouthCOMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: the Finnish Cultural Foundation, Central Finland Regional Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 21000039071
Record Dates: First submitted 2017-09-01; First posted 2017-09-07 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Well-being
Keywords: Adolescents; Web- and mobile-based intervention; Acceptance and Commitment therapy; Psychological well-being; Career preparation; Lifecontrol; Successful educational transitions; Learning difficulties; Psychological flexibility and mindfulness skills
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Treatment, Parallel assessment, Randomized, Efficacy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Face-to-face and online support group (Experimental): Behavioral: Structured web- and mobile-based intervention with Youth COMPASS program to support adolescents' well-being, career preparation and life-control and subsequently support successful transition to upper secondary education. The Youth COMPASS is the five-week online program according to principles of Acceptance and Commitment Therapy aiming to enhance adolescents' psychological flexibility by guiding adolescents in exploring their values and setting goals and changing behaviors according to their goals (week 1), and learning acceptance defusion and mindfulness skills (weeks 2-3) and integrating these skills into their personal life (weeks 4-5). The participants in this condition receive weekly online support and feedback from their individually assigned coach. In addition, they meet their coach twice in the face-to-face meetings. The aim of the meetings is to increase adolescents' internal motivation and thereby participation in the program.
  Interventions: Behavioral: Experimental: face-to-face and online support group:
- Only online support group (Experimental): Behavioral: web- and mobile-based intervention with Youth COMPASS program to support adolescents' well-being, career preparation and life-control and subsequently support successful transition to upper secondary education. The Youth COMPASS is a five-week online program according to principles of Acceptance and Commitment Therapy aiming to enhance adolescents' psychological flexibility by guiding adolescents in exploring their values and setting goals and changing behaviors according to their goals (week 1), and learning acceptance defusion and mindfulness skills (weeks 2-3) and integrating these skills into their personal life (weeks 4-5). The participants in this condition receive weekly online support and feedback from their individually assigned coach.
  Interventions: Behavioral: Experimental: only online support group:
- Control group (Experimental): Behavioral: No intervention, school counseling as usual
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Experimental: face-to-face and online support group: — 5-week intervention according to Acceptance and Commitment Therapy principles with the web-and mobile-based Youth COMPASS program, face-to-face support (2 meetings) and weekly online mobile support and feedback from the individually assigned coach (one third of the participants is randomly assigned to this group)
  Arms: Face-to-face and online support group
Behavioral: Experimental: only online support group: — 5-week intervention according to ACT principles with the web-and mobile-based Youth COMPASS program, no face-to-face support, weekly mobile online support and feedback from the individually assigned coach (one third of the participants is randomly assigned to this group)
  Arms: Only online support group
Behavioral: Control — Control group, no intervention, school counseling as usual. (one third of the participants is randomly assigned to this group)
  Arms: Control group

SUMMARY:
The aim of this randomized control trial is to examine effectiveness of individually tailored web- and mobile-based Acceptance- and Commitment Therapy interventions to promote adolescents' well-being and life-control and subsequently support their successful transition from basic education to upper secondary education. Our additional aim is to examine to what extent the effectiveness of the intervention varies according to intervention intensity and according to risk for school failure. The five-week structured intervention is delivered using the novel web-and mobile-based program Youth COMPASS following the principles of the Acceptance and Commitment Therapy (ACT). The Internet context is assumed to be particularly motivating for youth who enjoy spending time online using different social media. Internet-based interventions have several advantages; they can include more information and treatment components than traditionally delivered treatments and that intervention programs are accessible at any time and at any place. Another unique aspect of the Youth COMPASS is the fact that it is individually-tailored. Each participant have an individually assigned online coach who provides support and encouragement, reminds about Youth COMPASS, sends individualized feedback, and recommends different exercises. The study hypothetizes that the Youth COMPASS is more effective than school counseling as usual. More specifically, the Youth COMPASS is expected to be more effective when it is combined with face-to-face support than when support and feedback are provided only via the Internet. Also, the Youth COMPASS with no face-to-face support (online only) is expected to be more effective than receiving only regular school counseling. Finally, the Youth COMPASS is expected to be more effective for students at risk for school failure than for students without risk for school failure, especially when at risk-adolescents receive more intensive support (i.e., both online and face-to-face support).

DETAILED DESCRIPTION:
The aim of this randomized control trial is to examine effectiveness of individually tailored web- and mobile-based Acceptance- and Commitment Therapy interventions to promote adolescents' well-being and life-control and subsequently support their successful transition from basic education to upper secondary education. Our additional aim is to examine to what extent the effectiveness of the intervention varies according to intervention intensity and according to risk for school failure. The five-week structured intervention is delivered using the novel web-and mobile-based program Youth COMPASS following the principles of the Acceptance and Commitment Therapy (ACT). The Internet context is assumed to be particularly motivating for youth who enjoy spending time online using different social media. Internet-based interventions have several advantages; they can include more information and treatment components than traditionally delivered treatments and that intervention programs are accessible at any time and at any place. Another unique aspect of the Youth COMPASS is the fact that it is individually-tailored. Each participant have an individually assigned online coach who provides support and encouragement, reminds about Youth COMPASS, sends individualized feedback, and recommends different exercises. The study hypothetizes that the Youth COMPASS is more effective than school counseling as usual. More specifically, the Youth COMPASS is expected to be more effective when it is combined with face-to-face support than when support and feedback are provided only via the Internet. Also, the Youth COMPASS with no face-to-face support (online only) is expected to be more effective than receiving only regular school counseling. Finally, the Youth COMPASS is expected to be more effective for students at risk for school failure than for students without risk for school failure, especially when at risk-adolescents receive more intensive support (i.e., both online and face-to-face support). The participants of the effectiveness study of the Youth COMPASS are selected from the participants of the broader longitudinal STAIRWAY (TIKAPUU in Finnish) - From Primary School to Secondary School study, which follows a community sample of Finnish adolescents (n~850) across critical educational transitions. The overall aim of the STAIRWAY project is to broaden our understanding of the individual- and environment-related factors that promote learning, well-being and successful educational transitions.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents (n = 120) who have risk for school failure (learning difficulties or low grade point average without learning difficulties)
* Randomly chosen adolescents (n=120) from the same classrooms who have no risk for school failure

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 249 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Life satisfaction (Diener et al., 1985) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Self-esteem (Rosenberg, 1965), | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Depressive symptoms (Salokangas et al., 1995) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Stress (Elo et al., 2003) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Difficulties and Strenghts questionnaire (SDQ, Goodman et al. 1997) measuring emotional symptoms, hyperactivity, conduct problems and prosociality | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Well-being in school (World Health Organization) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Career choice preparedness (Koivisto et al., 2011) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Educational expectations | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.

SECONDARY OUTCOMES:
Psychological flexibility (Greco et al., 2008) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Mindfulness skills (Ciarrochi et al., 2011) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Identity formation (DIDS; Luyckx et al., 2008; see also Marttinen et al., 2016) | Change from baseline at 2, 6, 12 and 18 months after the intervention
  In addition to self-reports, also school register information is collected regarding academic performance, school absences and progress in studies.
Truancy | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
School grades | Four years from the baseline.
  In addition to self-reports, also school register information is collected.
Initiation of upper secondary education | Four years from the baseline.
  In addition to self-reports, also school register information is collected.
Progress in upper secondary studies | Four years from the baseline.
  In addition to self-reports, also school register information is collected.
Changes in study field in upper secondary education | Four years from the baseline.
  In addition to self-reports, also school register information is collected.
Staying in vs. dropping out of education | Four years from the baseline.
  In addition to self-reports, also school register information is collected.
Graduation time | Four years from the baseline.
  In addition to self-reports, also school register information is collected.

OTHER OUTCOMES:
Achievement strategies (Nurmi et al., 1995) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Academic buoyancy (Martin & Marsh, 2008) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Recovery from school work (see also Winwood et al., 2005) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Child-Parent relationship (Pianta, 1992) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Student-Teacher relationship (Pianta, 2001) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Best Friend-Student (Bukowski et al., 1994) relationship | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Temperament (Rothbart & Ellis, 2001) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Substance use (Rimpelä et al., 2003) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Loneliness (World Health Organization) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Health behaviors (World Health Organization) | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Dating | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.
Having hobbies | Change from baseline at 2, 6, 12 and 18 months after the intervention.
  Study has five timepoints when same questionnaires are administered to assess possible changes in the outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Noona Kiuru, PhD, Principal Investigator — Department of Psychology, University of Jyväskylä, Finland
Locations (1):
- Department of Psychology, University of Jyväskylä, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: Yes
Other researchers are encouraged to use the data; however, it requires a research plan and the permission of the research team. Also, at least one of the team members, who know the data well, should be a co-author in all the articles that are written from the data.
  After 10 years of the data collection, those parts of the data that are not too sensitive (e.g., part of the questionnaire data), will be prepared in collaboration with a Finnish Social Science data Archive in a format that is easily accessible for other researchers. However, using data requires a research plan and the permission of the research team. Also, at least one of the team members, who know the data well, should be a co-author in all the articles that are written from the data.